CLINICAL TRIAL: NCT00640822
Title: A Phase 3 Study Comparing an Ointment Containing Calcipotriol 25 mcg/g Plus Hydrocortisone 10 mg g With Tacalcitol 4 mcg/g Ointment and the Ointment Vehicle Alone, All Applied Once Daily in the Treatment of Psoriasis Vulgaris on the Face and on the Intertriginous Areas
Brief Title: Efficacy and Safety of Calcipotriol Plus Hydrocortisone Ointment Compared With Tacalcitol Ointment in Patients With Psoriasis on the Face and Skin Folds
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LEO 80190-O22
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Results first posted 2010-12-21 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2015-04

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — calcipotriene

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Calcipotriol plus Hydrocortisone ointment (Experimental): Calcipotriol plus Hydrocortisone ointment once daily for up to 8 weeks
  Interventions: Drug: Calcipotriol plus hydrocortisone ointment
- Tacalcitol (Active Comparator): Tacalcitol once daily for up to 8 weeks
  Interventions: Drug: Tacalcitol Ointment
- Calcipotriol plus Hydrocortisone ointment vehicle (Placebo Comparator): Calcipotriol plus Hydrocortisone ointment vehicle once daily for up to 8 weeks
  Interventions: Drug: Calcipotriol plus hydrocortisone ointment vehicle

INTERVENTIONS:
Drug: Calcipotriol plus hydrocortisone ointment vehicle — Once daily application for up to 8 weeks
  Arms: Calcipotriol plus Hydrocortisone ointment vehicle
Drug: Tacalcitol Ointment — Once daily application for up to 8 weeks
  Arms: Tacalcitol
Drug: Calcipotriol plus hydrocortisone ointment — Once daily application for up to 8 weeks
  Arms: Calcipotriol plus Hydrocortisone ointment

SUMMARY:
There are few therapies suitable for the treatment of psoriasis on the face and skin folds. As these areas are sensitive, irritation and other adverse reactions are more common than elsewhere on the body. The purpose of the study is to compare the efficacy and safety of once daily treatment for up to 8 weeks of an ointment containing calcipotriol 25 mcg/g plus hydrocortisone 10 mg/g with tacalcitol 4 mcg/g ointment and the ointment vehicle alone in patients with psoriasis vulgaris on the face and on the intertriginous ares

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of psoriasis vulgaris involving the face
* Clinical signs of psoriasis vulgaris on the trunk and/or the limbs, or earlier diagnosed with psoriasis vulgaris on the trunk and/or the limbs
* An extent of psoriatic involvement of the face of at least 10 cm2 (the sum of all facial lesions)
* Treatment areas (the face and the intertriginous areas) amenable to topical treatment with a maximum of 10 g of ointment per day
* Disease severity graded as mild, moderate, severe or very severe according to the investigator's global assessment of disease severity of the face

Exclusion Criteria:

* Systemic treatments with all other therapies than biologicals, with a potential effect on psoriasis vulgaris (e.g., corticosteroids, vitamin D analogues, retinoids, immunosuppressants) within the 4-week period prior to randomisation
* Systemic use of biological treatments, whether marketed or not, directed against or with a potential effect on psoriasis vulgaris (e.g., alefacept, efalizumab, etanercept, infliximab, adalimumab) within 3 months prior to randomisation
* PUVA therapy or Grenz ray therapy within the 4-week period prior to randomisation
* UVB therapy within the 2-week period prior to randomisation
* Topical treatment of the face and the intertriginous areas within the 2-week period prior to randomisation (use of emollients is allowed on treatment areas during this 2-week period, but not during the study)
* Topical treatment with very potent WHO group IV corticosteroids within the 2-week period prior to randomisation
* Initiation of or expected changes in concomitant medication that may affect psoriasis vulgaris (e.g., beta blockers, anti-malaria drugs, lithium and ACE inhibitors) during the study
* Systemic treatment with vitamin D preparations above 500 IU per day
* Current diagnosis of erythrodermic, exfoliative, guttate or pustular psoriasis
* Patients with any of the following conditions present on the treatment area: viral (e.g., herpes or varicella) lesions of the skin, fungal and bacterial skin infections, parasitic infections, skin manifestations in relation to syphilis or tuberculosis, rosacea, perioral dermatitis, acne vulgaris, atrophic skin, striae atrophicae, fragility of skin veins, ichthyosis, acne rosacea, ulcers and wounds
* Other inflammatory skin diseases (e.g., seborrhoeic dermatitis, contact dermatitis and cutaneous mycosis) that may confound the evaluation of psoriasis vulgaris on the face or on the intertriginous areas
* Planned exposure to sun, UVA or UVB that may affect the psoriasis vulgaris during the study
* Known or suspected severe renal insufficiency or severe hepatic disorders
* Known or suspected disorders of calcium metabolism associated with hypercalcemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 782 (Actual)
Dates: Start 2008-02; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Fleming, MD, Principal Investigator — Ninewells Hospital & Medical School
Locations (3):
- Probity Medical Research, Waterloo, Ontario, Canada
- Hôpital de l'Archet, Nice, France
- Ninewells Hospital & Medical School, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first subject visit was 5 Mar 2008. Date of last subject visit was 18 Jun 2009. Patients came from hospital outpatient clinics or private practice
Pre-assignment Details: Forty-one subjects were not randomised. Most we screen failures or did not have the required extent of disease or withdrew before randomization
Groups:
- Tacalcitol Ointment: Tacalcitol once daily for up to 8 weeks
Period: Overall Study
Arm/Group | Calcipotriol Plus Hydrocortisone Ointment | Tacalcitol Ointment | Calcipotriol Plus Hydrocortisone Ointment Vehicle
Started | 322 | 317 | 102
Completed | 279 | 258 | 77
Not Completed | 43 | 59 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcipotriol Plus Hydrocortisone Ointment | Tacalcitol Ointment | Calcipotriol Plus Hydrocortisone Ointment Vehicle | Total
Number analyzed (Participants) | 322 | 317 | 102 | 741
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (15.5) | 49 (15.5) | 48.8 (14.2) | 48.5 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 136 | 41 | 303
  Male | 196 | 181 | 61 | 438
Region of Enrollment [Number; unit: participants]
  France | 95 | 83 | 38 | 216
  Canada | 131 | 129 | 37 | 297
  United Kingdom | 96 | 105 | 27 | 228

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Controlled Disease According to the Investigator Assessment of the Face at Week 8
Time Frame: Week 8
Measure: Number; unit: Participants
Arm/Group | Calcipotriol Plus Hydrocortisone Ointment | Tacalcitol Ointment | Calcipotriol Plus Hydrocortisone Ointment Vehicle
Number analyzed (Participants) | 322 | 317 | 102
Participants | 183 | 147 | 37

2. Secondary Outcome: Overall Disease Severity of the Face According to the Investigator's Assessment
Time Frame: Week 4
Reporting Status: Not Posted

3. Secondary Outcome: Total Sign Score of the Face
Time Frame: Week 8
Reporting Status: Not Posted

4. Secondary Outcome: Severity Scores for Redness, Thickness and Scaliness of the Face
Time Frame: Week 8
Reporting Status: Not Posted

5. Secondary Outcome: Overall Disease Severity of the Intertriginous Areas According to the Investigator's Assessment
Time Frame: Week 8
Reporting Status: Not Posted

6. Secondary Outcome: Total Sign Score of the Intertriginous Areas
Time Frame: Week 8
Reporting Status: Not Posted

7. Secondary Outcome: Patients With Relapse During the Study and Time to Relapse
Time Frame: Week 8-16
Reporting Status: Not Posted

8. Secondary Outcome: Patients With Rebound During the Study
Time Frame: Week 8-16
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: The safety analysis set consists of all randomised subjects who received any treatment with trial medication and for whom the presence or confirmed absence of adverse events was available. Two subjects withdrew within the first week of the study and did not apply any study medication so they were excluded from the safety analysis set.
Arm/Group | Calcipotriol Plus Hydrocortisone Ointment | Tacalcitol Ointment | Calcipotriol Plus Hydrocortisone Ointment Vehicle
Serious Adverse Events (participants affected / at risk) | 5/321 | 3/316 | 4/102
Other Adverse Events (participants affected / at risk) | 13/321 | 30/316 | 2/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Calcipotriol Plus Hydrocortisone Ointment (N=321) | Tacalcitol Ointment (N=316) | Calcipotriol Plus Hydrocortisone Ointment Vehicle (N=102)
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Calcipotriol Plus Hydrocortisone Ointment (N=321) | Tacalcitol Ointment (N=316) | Calcipotriol Plus Hydrocortisone Ointment Vehicle (N=102)
Erythema (Skin and subcutaneous tissue disorders) | 13 | 30 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Company acknowledges the investigators right to publish the entire results of the study, irrespective of outcome. The Company retains the right to have any publication submitted to the Company for review at least 30 days prior to the same paper being submitted for publication or presentation. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.